CLINICAL TRIAL: NCT00349336
Title: A Randomized, Open Label Trial to Assess the Steady State Pharmacokinetics of Avastin Given With Either XELOX or FOLFOX-4 in Patients With Metastatic Colorectal Cancer
Brief Title: A Study of Avastin (Bevacizumab) in Combination With XELOX or FOLFOX-4 in Patients With Metastatic Colorectal Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO20254
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Results first posted 2010-02-26 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; XELOX; Folfox protocol

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: XELOX
- 2 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: FOLFOX-4

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 7.5mg/kg iv on day 1 of each 3 week cycle
  Arms: 1
Drug: XELOX — As prescribed
  Arms: 1
Drug: bevacizumab [Avastin] — 5mg/kg iv on day 1 of each 2 week cycle
  Arms: 2
Drug: FOLFOX-4 — As prescribed
  Arms: 2

SUMMARY:
This 2 arm study will compare the pharmacokinetics and safety of Avastin at steady state under 2 different dosing regimens, in combination with XELOX (oxaliplatin + Xeloda) or FOLFOX-4 (oxaliplatin, leucovorin and 5-fluorouracil). Patients randomized to the XELOX arm will receive Avastin (7.5mg/kg iv) on Day 1 of each 3 week cycle; patients randomized to the FOLFOX-4 arm will receive Avastin (5mg/kg iv) on Day 1 of each 2 week cycle. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* adenocarcinoma of the colon or rectum, with metastatic or locally advanced disease;
* >=1 target lesion.

Exclusion Criteria:

* patients who have previously received systemic treatment for advanced or metastatic disease;
* patients who have received adjuvant treatment for non-metastatic disease in past 3 months;
* previous therapy with oxaliplatin or Avastin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Australia (3):
  - Box Hill
  - Fitzroy
  - Sydney
- Canada (3):
  - Brampton, Ontario
  - Hamilton, Ontario
  - Toronto, Ontario
- Christchurch, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 64 patients in 7 centers were enrolled between 01 August 2006 to 28 May 2008. 37 were included in the pharmacokinetic (PK) analyses.
Groups:
- XELOX+Bevacizumab: XELOX regimen = oxaliplatin in combination with capecitabine. Bevacizumab 7.5 mg/kg IV followed by oxaliplatin 130 mg/m² IV on Day 1 in combination with capecitabine, administered orally at a dose of 1000 mg/m² twice daily (BID); 3-week cycles up to 48 weeks (Cycle 16).
- FOLFOX-4+Bevacizumab: FOLFOX-4 regimen = oxaliplatin in combination with infusional 5-fluorouracil and leucovorin. Bevacizumab 5.0 mg/kg IV followed by oxaliplatin 85 mg/m² IV on Day 1 concomitantly with leucovorin 200 mg/m² IV, followed by 5-fluorouracil administered as a 400 mg/m² bolus injection, and then as a 600 mg/m² continuous infusion on Days 1 and 2; 2-week cycles for up to 48 weeks (Cycle 24).
Period: Overall Study
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Started | 32 | 32
Completed | 19 | 18
Not Completed | 13 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab | Total
Number analyzed (Participants) | 32 | 32 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 55.9 (12.56) | 57.9 (10.84) | 56.9 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 19 | 15 | 34

OUTCOME MEASURES:

1. Secondary Outcome: Time Zero to Last Measurable Plasma Concentration of Bevacizumab
Description: Area under the serum concentration-time curve from time zero to the time of the last measurable plasma concentration (AUC 0-last). Estimation of the parameter was performed using non-compartmental methods.
Time Frame: Up to 48 weeks
Population: 42 patients participated in pharmacokinetic (PK) assessments and of those, 37 were included in the PK analysis. Two patients receiving XELOX+BV were not included in the PK analysis due to protocol violations.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Number analyzed (Participants) | 19 | 18
day*ug/mL | 2457.19 (359.5) | 1709.8 (497.0)

2. Primary Outcome: Weekly Steady-state Exposure of Bevacizumab
Description: Area under the serum concentration-time curve per week, at steady state (AUCss per week). Estimation of the parameter was performed using non-compartmental methods.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Number analyzed (Participants) | 19 | 18
day*ug/mL | 4090.3 (1047.6) | 4022.4 (1774.2)

3. Secondary Outcome: Steady-state Exposure of Bevacizumab From Time Zero to Tau
Description: Area under the serum concentration-time curve from time zero to tau, at steady state (AUCss 0-tau), where tau was the length of the cycle, i.e., tau = 3 weeks for XELOX+BV and tau = 2 weeks for FOLFOX-4+BEV. Estimation of the parameter was performed using non-compartmental methods.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Number analyzed (Participants) | 19 | 18
day*ug/mL | 2457.0 (360.6) | 1758.4 (468.5)

4. Secondary Outcome: Maximum Serum Concentration of Bevacizumab at Steady State
Description: Maximum serum concentration at steady state (Css,max). Estimation of the parameter was performed using non-compartmental methods.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Number analyzed (Participants) | 19 | 18
ug/mL | 242 (31.6) | 215.6 (53.2)

5. Secondary Outcome: Minimum Serum Concentration of Bevacizumab at Steady State
Description: Minimum serum concentration at steady state (Css, min). Estimation of the parameter was performed using non-compartmental methods.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Number analyzed (Participants) | 19 | 18
ug/ml | 59.6 (14.1) | 80.0 (25.5)

6. Secondary Outcome: Serum Clearance of Bevacizumab
Description: Serum clearance (CL). Estimation of the parameter was performed using non-compartmental methods.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Number analyzed (Participants) | 19 | 18
L/day | 0.236 (0.051) | 0.226 (0.056)

7. Secondary Outcome: Time of Maximum Serum Concentration of Bevacizumab
Description: Time of maximum serum concentration (tmax). Estimation of the parameter was performed using non-compartmental methods.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Number analyzed (Participants) | 19 | 18
hr | 6.442 (6.786) | 4.958 (3.596)

8. Secondary Outcome: Volume of Distribution of Bevacizumab at Steady State
Description: Volume of distribution at steady state (Vss). Estimation of the parameter was performed using non-compartmental methods.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Number analyzed (Participants) | 19 | 18
L | 4.932 (1.409) | 4.908 (1.563)

9. Secondary Outcome: Terminal Half-life of Bevacizumab
Description: Terminal half-life (t1/2) (apparent elimination half-life). Estimation of the parameter was performed using non-compartmental methods.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Number analyzed (Participants) | 19 | 18
hr | 381.2 (91.7) | 394.1 (121.8)

ADVERSE EVENTS:
Arm/Group | XELOX+Bevacizumab | FOLFOX-4+Bevacizumab
Serious Adverse Events (participants affected / at risk) | 9/32 | 15/32
Other Adverse Events (participants affected / at risk) | 32/32 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XELOX+Bevacizumab (N=32) | FOLFOX-4+Bevacizumab (N=32)
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Rectal Haemorhage (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 1
Catheter Thrombosis (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Anorectal Infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2
Bile Duct Obstruction (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XELOX+Bevacizumab (N=32) | FOLFOX-4+Bevacizumab (N=32)
Diarrhoea (Gastrointestinal disorders) | 20 | 23
Nausea (Gastrointestinal disorders) | 26 | 16
Abdominal Pain (Gastrointestinal disorders) | 11 | 8
Constipation (Gastrointestinal disorders) | 10 | 9
Vomiting (Gastrointestinal disorders) | 8 | 9
Stomatitis (Gastrointestinal disorders) | 5 | 7
Flatulence (Gastrointestinal disorders) | 9 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 5
Haemorrhoids (Gastrointestinal disorders) | 3 | 3
Abdominal Distension (Gastrointestinal disorders) | 3 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 2 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 4
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 2
Oral Pain (Gastrointestinal disorders) | 1 | 2
Anal Fissure (Gastrointestinal disorders) | 0 | 2
Anorectal Discomfort (Gastrointestinal disorders) | 0 | 2
Gingival Bleeding (Gastrointestinal disorders) | 2 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 2
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 2
Mouth Ulceration (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 24 | 23
Temperature Intolerance (General disorders) | 15 | 12
Mucosal Inflammation (General disorders) | 6 | 11
Pyrexia (General disorders) | 3 | 7
Oedema Peripheral (General disorders) | 1 | 6
Influenza Like Illness (General disorders) | 2 | 3
Injection Site Discolouration (General disorders) | 3 | 2
Pain (General disorders) | 3 | 2
Chest Pain (General disorders) | 2 | 2
Chills (General disorders) | 1 | 2
Mucosal Haemorrhage (General disorders) | 2 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 15 | 16
Neuropathy Peripheral (Nervous system disorders) | 15 | 15
Headache (Nervous system disorders) | 10 | 10
Dizziness (Nervous system disorders) | 6 | 6
Paraesthesia (Nervous system disorders) | 4 | 7
Dysgeusia (Nervous system disorders) | 3 | 4
Dysaesthesia (Nervous system disorders) | 1 | 2
Cranial Neuropathy (Nervous system disorders) | 2 | 0
Disturbance in Attention (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 2
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 18 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 9
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 | 7
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 3
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 4 | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Skin Discolouration (Skin and subcutaneous tissue disorders) | 3 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal Ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 3
Groin Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Rhinitis (Infections and infestations) | 5 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 4
Nasopharyngitis (Infections and infestations) | 2 | 2
Oral Herpes (Infections and infestations) | 2 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 3
Central Line Infection (Infections and infestations) | 0 | 2
Eye Infection (Infections and infestations) | 2 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 2
Tooth Infection (Infections and infestations) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 16 | 8
Decrease Appetite (Metabolism and nutrition disorders) | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypertension (Vascular disorders) | 7 | 7
Thrombosis (Vascular disorders) | 1 | 4
Flushing (Vascular disorders) | 0 | 3
Hot Flush (Vascular disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 4 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 9 | 9
Eye Pain (Eye disorders) | 3 | 2
Lacrimation Increased (Eye disorders) | 0 | 5
Weight Decreased (Investigations) | 1 | 5
Gamma-Glutamyltransferase Increased (Investigations) | 2 | 1
Hypersensitivity (Immune system disorders) | 0 | 4
Proteinuria (Renal and urinary disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.